CLINICAL TRIAL: NCT00453401
Title: The Safety, Pharmacokinetics, and Efficacy of NB-001 (0.1%, 0.3%, 0.5%) in Subjects With Recurrent Herpes Labialis
Brief Title: Safety, Pharmacokinetics, and Efficacy Study of NB-001 to Treat Recurrent Herpes Labialis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NanoBio Corporation (Industry)
Responsible Party: Mary Flack, MD, NanoBio Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB-001-003
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Herpes Labialis
Keywords: cold sore
MeSH Terms: conditions — Herpes Labialis | interventions — 5-((2-(6-Amino-9H-purin-9-yl) ethyl) amino)-1-pentanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: NB-001

SUMMARY:
Purpose of this study is to determine the safety and efficacy of topical applications of NB-001 as compared to placebo for the treatment of recurrent herpes labialis.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age of either gender
* Good general health
* History of recurrent herpes labialis with at least 3 episodes per year

Exclusion Criteria:

* Pregnant and/or nursing female
* Lesions or irritation on or around the lips that would interfere with recognition of a herpes labialis attack
* Treatment with topical steroids, antivirals, or new topical products on or around the lips in the week prior to the onset of an attack
* Known allergies to topical creams, ointments or medications.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Time to healing as assessed by the subject.

SECONDARY OUTCOMES:
Percent of subjects with healing by days 3, 4,and 5 as assessed by the subject.

CONTACTS AND LOCATIONS:
Overall Officials: William Abramovits, MD, Principal Investigator — Dermatology Treatment and Research Center; Jeffrey Adelglass, MD, Principal Investigator — Research Across America; Maurice Archuleta, MD, Principal Investigator — Front Range Clinical Research; Brian Bock, DO, Principal Investigator — Bock Clinical Research Incorporated; Alicia Bucko, DO, Principal Investigator — Academic Dermatology Associates; Teresa Coats, MD, Principal Investigator — Benchmark Research; Lisa Cohen, DO, Principal Investigator — Suncoast Clinical Research; John Eck, MD, Principal Investigator — Advanced Clinical Research Incorporated; Douglass Forsha, MD, Principal Investigator — South Valley Dermatology Center; David Fried, MD, Principal Investigator — Omega Medical Research; Helen Henry, MD, Principal Investigator — Westover Heights Clinic; Michael T Jarratt, MD, Principal Investigator — Derm Research Incorporated; Terry Jones, MD, Principal Investigator — J & S Studies; Steven Kaster, MD, Principal Investigator — Wenatchee Valley Medical Center; Leon Kircik, MD, Principal Investigator — DermResearch, PLCC; Ronica Kluge, MD, Principal Investigator — Clinical Physiology Associates; Elias Kolettis, MD, Principal Investigator — Clinical Research of West Florida; Oswald Mikell, MD, Principal Investigator — Okati Research Center, LLC; Eugene Monroe, MD, Principal Investigator — Advance Healthcare; Edward Pornoy, MD, Principal Investigator — Westlake Medical Research; Harvey Resnick, MD, Principal Investigator — R/D Clinical Research Incorporated; Dennis Riff, MD, Principal Investigator — Advanced Clinical Research Institute; Mark A Ringold, MD, Principal Investigator — New River Valley Research Institute; Ronald Savin, MD, Principal Investigator — PC; Daniel Stewart, MD, Principal Investigator — MI Center for Skin Care Research; Cynthia B Strout, MD, Principal Investigator — Coastal Carolina Research Center; Wayne Harper, MD, Principal Investigator — Wake Research Associates, LLM; Timothy Howard, MD, Principal Investigator — Medical Affiliated Reseach Center Incorporated
Locations (28):
- United States (28):
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Advanced Clinical Research Institute, Anaheim, California
  - Westlake Medical Research, Westlake Village, California
  - Front Range Clinical Research, Wheat Ridge, Colorado
  - The Savin Center, PC, New Haven, Connecticut
  - Clinical Research of West Florida, Clearwater, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Advanced Clinical Research, Inc., Boise, Idaho
  - DermResearch, PLCC, Louisville, Kentucky
  - MI Center for Skin Care Research, Clinton Township, Michigan
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Wake Research Associates, LLM, Raleigh, North Carolina
  - Westover Heights Clinic, Portland, Oregon
  - Lederach Family Medicine, Harleysville, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Okatie Research Center, LLC, Beaufort, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Benchmark Research, Austin, Texas
  - DermResearch Inc., Austin, Texas
  - J&S Studies Inc., Bryan, Texas
  - Dermatology Treatment & Research Center, Dallas, Texas
  - Research Across America, Dallas, Texas
  - R/D Clinical Research, Inc, Lake Jackson, Texas
  - South Valley Dermatology Center, West Jordan, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Advanced Healthcare, Milwaukee, Wisconsin